CLINICAL TRIAL: NCT00301444
Title: A Pilot Study to Assess the Efficacy of Mirror-Box and Mental Visualization Treatments on Phantom Limb Pain
Brief Title: A Study to Test the Effectiveness of Mirror-Box and Mental Visualization Treatments on Phantom Limb Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Department of Defense (U.S. Federal Agency)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DCI P05-A008
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-04

CONDITIONS: Amputation; Phantom Limb; Pain
Keywords: phantom limb pain; limb amputation
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: mirror-box treatment
Behavioral: Mental visualization

SUMMARY:
The researchers propose to conduct a pilot study on the efficacy of mirror-box and mental visualization treatments on phantom limb pain. The trial will last for 4 months and during the first month, data will be gathered daily on the number of episodes of phantom limb pain, the average length of episodes, average intensity of pain, and worst intensity of pain. In addition, the rapidity of pain relief, the length of therapy needed to sustain long-lasting pain relief, and whether use of these two treatment methods during rehabilitation can provide sustained and/or permanent pain relief will be determined. Cognitive testing will also be performed to determine the effect of limb amputation on cognition and mood with results being compared to an on-going study of similar effects in patients with chronic (> 3 months) limb amputation.

The inclusion of subjects with phantom limb pain in upper extremity amputations has recently been approved.

DETAILED DESCRIPTION:
A total of forty-eight (48) subjects with be enrolled - twenty-four (24) with any unilateral lower limb amputation and twenty-four (24) with any unilateral upper limb amputation. Subjects will be randomized for assignment into three treatment conditions: eight (8) lower and eight (8) upper limb subjects (50% with left-sided amputations) will use mental visualization of foot or hand movements, eight (8) lower and eight (8) upper limb subjects (50% with left-sided amputations) will use an open mirror- box to visualize the reflected image of their intact foot or hand, and eight (8) lower and eight (8) upper limb subjects (50% with left-sided amputations) will use a closed mirror- box (unable to visualize a reflected image). Subjects will use their assigned therapy for 20 minutes daily. Subjects using the closed mirror-box or mental visualization treatments will be switched to mirror therapy if they have not significantly improved following 4 weeks. The subjects for this study will be recruited from the Walter Reed Army Medical Center Amputee clinic. Up to sixty (60) subjects will be recruited and screened according to the inclusion and exclusion criteria since we expect that some may not qualify or drop-out sooner than the scheduled 4-month completion time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 70 years of age, active duty military, beneficiary, or retiree.
* Written informed consent and written authorization for use or release of health and research study information.
* Any single unilateral upper or lower limb amputation with the presence of phantom limb pain.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Normal neurological examination.
* Degree of pain evaluated by VAS scoring a minimum of 3 cm at time of screening for entry into the study, with a minimum of three episodes per week.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* Age less than 18 or greater than 70.
* Bilateral upper or lower limb amputation.
* Presence of traumatic brain injury - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening which is currently performed routinely on patients by the TBI program at WRAMC and noted in the patient's medical record.
* Known uncontrolled systemic disease- known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Concurrent participation in another investigational drug or device study for phantom limb pain or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study.
* Subjects with lack of effort as determined by the neurologist or physiatrist. Subjects will be screened for effort using the Test of Memory Malingering (TOMM) first in order to exclude those with blatant exaggeration or malingering.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-03; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Significant decrease in the level of phantom limb pain at 4 weeks.

SECONDARY OUTCOMES:
Significant decrease in the number and duration of daily phantom limb pain episodes at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jack W Tsao, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Carlen PL, Wall PD, Nadvorna H, Steinbach T. Phantom limbs and related phenomena in recent traumatic amputations. Neurology. 1978 Mar;28(3):211-7. doi: 10.1212/wnl.28.3.211. PMID 564474
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] MacLachlan M, McDonald D, Waloch J. Mirror treatment of lower limb phantom pain: a case study. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):901-4. doi: 10.1080/09638280410001708913. PMID 15497919
- [Background] Jackson PL, Lafleur MF, Malouin F, Richards CL, Doyon J. Functional cerebral reorganization following motor sequence learning through mental practice with motor imagery. Neuroimage. 2003 Oct;20(2):1171-80. doi: 10.1016/S1053-8119(03)00369-0. PMID 14568486
- [Background] Ramachandran VS, Altschuler EL, Stone L, Al-Aboudi M, Schwartz E, Siva N. Can mirrors alleviate visual hemineglect? Med Hypotheses. 1999 Apr;52(4):303-5. doi: 10.1054/mehy.1997.0651. PMID 10465667
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Ochipa C, Rapcsak SZ, Maher LM, Rothi LJ, Bowers D, Heilman KM. Selective deficit of praxis imagery in ideomotor apraxia. Neurology. 1997 Aug;49(2):474-80. doi: 10.1212/wnl.49.2.474. PMID 9270580
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Katz J, Melzack R. Pain 'memories' in phantom limbs: review and clinical observations. Pain. 1990 Dec;43(3):319-336. doi: 10.1016/0304-3959(90)90029-D. PMID 2293143
- [Derived] Finn SB, Perry BN, Clasing JE, Walters LS, Jarzombek SL, Curran S, Rouhanian M, Keszler MS, Hussey-Andersen LK, Weeks SR, Pasquina PF, Tsao JW. A Randomized, Controlled Trial of Mirror Therapy for Upper Extremity Phantom Limb Pain in Male Amputees. Front Neurol. 2017 Jul 7;8:267. doi: 10.3389/fneur.2017.00267. eCollection 2017. PMID 28736545